CLINICAL TRIAL: NCT01516320
Title: Mechanisms of Diabetes Relapse After Bariatric Surgery
Acronym: LAF26
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Blandine Laferrere (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Blandine Laferrere, Professor of Medicine, Columbia University, Columbia University
Organization: Columbia University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AAAO1101; R01DK067561 (NIH)
Record Dates: First submitted 2012-01-19; First posted 2012-01-24 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Gastric Bypass; Laparoscopic Banding; Vertical Sleeve Gastrectomy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gastric Bypass (GBP) Subjects (Experimental): Subjects enrolled in the study who are receiving Roux-en-Y Gastric Bypass surgical technique for treatment of their obesity.
  Interventions: Procedure: Roux-en-Y Gastric Bypass
- Laparoscopic adjustable gastric banding (LAGB) Subjects (Active Comparator): Subjects enrolled in the study who are receiving laparoscopic adjustable gastric banding surgical technique for treatment of their obesity.
  Interventions: Procedure: Laparoscopic adjustable gastric banding
- Vertical Sleeve Gastrectomy (VSG) Subjects (Active Comparator): Subjects enrolled in the study who are receiving vertical sleeve gastrectomy surgical technique for treatment of their obesity.
  Interventions: Procedure: Vertical Sleeve Gastrectomy

INTERVENTIONS:
Procedure: Roux-en-Y Gastric Bypass — A surgical technique in which the stomach is stapled into a smaller pouch and then attached directly to the small intestine, bypassing the rest of the original stomach. The goal of the surgery is weight loss.
  Arms: Gastric Bypass (GBP) Subjects
Procedure: Laparoscopic adjustable gastric banding — A surgical technique in which an inflatable silicone device placed around the top portion of the stomach, creating a smaller gastric pouch. The goal of the surgery is weight loss.
  Arms: Laparoscopic adjustable gastric banding (LAGB) Subjects
Procedure: Vertical Sleeve Gastrectomy — A surgical technique in which a large portion of the stomach is removed, leaving only a smaller gastric pouch. The goal of the surgery is weight loss.
  Arms: Vertical Sleeve Gastrectomy (VSG) Subjects

SUMMARY:
The objective of this study is to investigate the different mechanisms by which Gastric Bypass (GBP), laparoscopic adjustable gastric banding (LAGB) and vertical sleeve gastrectomy (VSG) affect glucose control. We wish to understand the role of weight loss versus changes in gut peptides in the short and long term in morbidly obese patients with Type 2 Diabetes Mellitus after GBP, LAGB or VSG. The 2 surgical groups will be compared at 10% equivalent weight loss and at after surgery in terms of gut hormones levels, insulin secretion and glucose control.

DETAILED DESCRIPTION:
The mechanisms of type 2 diabetes (T2DM) remission after gastric bypass surgery (GBP) are unclear. The levels of the gut hormones incretins and their effect on insulin secretion, which is impaired in T2DM, markedly increase after GBP. The anatomical changes of GBP, rather than weight loss, seem to be responsible for the changes of incretins. The objective of this proposal is to investigate the different mechanisms by which GBP, laparoscopic adjustable gastric banding (LAGB) and vertical sleeve gastrectomy (VSG) affect glucose control. We wish to understand the role of weight loss versus changes in gut peptides in the short and long term in morbidly patients with T2DM after GBP, LAGB or VSG.

AIM 1: Will study the short term changes of incretins levels and effect in obese individuals with T2DM after GBP, LAGB or VSG, before and 1 month after GBP or before and after equivalent weight loss after LAGB or VSG.

AIM 2: Will study the long-term (12 and 24 months after surgery) changes in the incretin effect on insulin secretion, in patients with T2DM after GBP, LAGB or VSG.

AIM 3: Will study the changes of insulin secretion to IV glucose (AIRg) and insulin sensitivity (Si), measured by the minimal model, in patients with T2DM after GBP, VSG or LAGB, before and at 24 months after the surgery, at weight stability under condition of controlled diet.

ELIGIBILITY:
Inclusion Criteria: Post GBP, LAGB or VSG Subjects

* Must be able to attend 4 study visits at St. Luke's Roosevelt Hospital Center in Manhattan, New York City
* History of Type 2 Diabetes before surgery

Inclusion Criteria:

* 35 < BMI < 50
* Non-Smoker
* Total Body Weight < 300 LBS
* 30<Age<60
* HbA1c < 9%
* Resting Blood Pressure < 160/100 mmHg
* Beta Blockers discontinued 2 weeks prior
* Fasting Triglyceride Concentration < 600 mg/dl (patient can be on dyslipidemia medications)
* Without recent (within last 6 months) CHD history (prior history of angioplasty or coronary artery bypass surgery with normal stress test ok)

Exclusion Criteria:

1. Patients with abnormal thyroid, renal function, known malabsorption syndrome or a seizure disorder requiring anti epileptic therapy, and/or elevation of liver enzymes three times above the normal limit.
2. Patients should not have significant secondary complications from diabetes that would preclude undergoing gastric by-pass surgery. This would include significant psychiatric, renal or neurological, or known active coronary artery disease.
3. Any abnormality during the maximum exercise stress test that indicates it would be unsafe to undergo bariatric surgery.
4. Currently pregnant or nursing.
5. Known cardiovascular disease
6. Patient with current mucosal (gastrointestinal, respiratory, urogenital) or skin (cellulitis) infection
7. HbA1c >9% and diabetes diagnosed more than 6 years prior to enrollment, or patients taking insulin or TZD (Avandia, Actos, Exenatide, DPP-IV inhibitors etc.) at the time of enrollment.
8. Patients diagnosed with intestinal conditions such as chronic diarrhea, diverticulitis, or irritable bowel syndrome. These clinical conditions would interfere with the collection and interpretation of the H2 breath test.
9. Any other condition which, in the opinion of the investigators, may make the candidate unsuitable for participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-05-13 (Actual); Primary Completion 2014-09-01 (Actual); Study Completion 2014-09-01 (Actual)

PRIMARY OUTCOMES:
Difference in insulin secretion between groups. | 0 - 48 months after surgery
  The investigators will assess insulin secretion in response to oral and intravenous nutrient and hormonal stimuli in the three groups.

SECONDARY OUTCOMES:
Difference in Incretin hormone response between groups. | 0 - 48 months after surgery
  The investigators will assess the endogenous incretin response to oral glucose stimulus after GBP.
Difference in Body composition between groups | 0 - 48 months after surgery
  The investigators will assess body composition (fat mass and fat distribution) in the 3 groups.

CONTACTS AND LOCATIONS:
Overall Officials: Blandine Laferrere, MD, Principal Investigator — New York Obesity Nutrition Research Center
Locations (1):
- New York Obesity Nutrition Research Center, St. Luke's-Roosevelt Hospital Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: New York Obesity Nutrition Research Center — http://www.nyorc.org/